CLINICAL TRIAL: NCT05045105
Title: Timing of Invasive Intracranial Pressure Monitoring Between Neurosurgeons and Intensive Care Physicians
Acronym: TIMING-ICP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Dr. Frank Rasulo, Associate Professor in Anesthesiology and Intensive Care, Università degli Studi di Brescia
Other Study IDs: NP4628
Record Dates: First submitted 2021-07-22; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Intracranial Hypertension; Timing of Invasive Intracranial Pressure Monitoring
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU physicians: Intensive Care physicians who will apply the method of invasive insertion of the intracerebral catheter for ICP monitoring
  Interventions: Other: Time necessary for ICP catheter placement by Intensive Care Physician vs Neurosurgeon following indication
- Neurosurgeons: Neurosurgeons who will apply the method of invasive insertion of the intracerebral catheter for ICP monitoring
  Interventions: Other: Time necessary for ICP catheter placement by Intensive Care Physician vs Neurosurgeon following indication

INTERVENTIONS:
Other: Time necessary for ICP catheter placement by Intensive Care Physician vs Neurosurgeon following indication — Time necessary for ICP catheter placement by Intensive Care Physician vs Neurosurgeon following indication and complications related to the maneuver between the two cohorts will be evaluated and compared.
  Other Names: Complications related to the maneuver between the two cohorts

SUMMARY:
Invasive intracranial pressure monitoring takes on essential importance in patients with traumatic brain injury and in all cerebral pathologies in which intracranial hypertension is the main cause of death.

Prolonged Intracranial Hypertension has been related to poor outcome and its occurrence has therefore to be assessed as soon as possible.

Invasive intracranial pressure monitoring performed by placing an intracerebral catheter is currently the gold standard technique for continuous ICP invasive monitoring. This maneuver has usually been performed by neurosurgeons, but recently this procedure has more often been carried out by intensivists, at the bedside.

Management of intracranial pressure handling and treatment is currently achieved by joint decisions between neurosurgeons and intensive care physicians, but differences in logistic matters and in the executive availability could impact on the dose of intracranial pressure to which patient is exposed.

The aim of this study is to compare timing of invasive intracranial pressure monitoring placement performed by intensive care physicians and neurosurgeons and to detect possible differences in the incidence of complications between the two groups.

DETAILED DESCRIPTION:
This perspective, multicentric and observational study will enroll patients at risk for developing intracranial hypertension, for whom it is thought invasive ICP monitoring is crucial for achieving the most appropriate treatment.

Indication to invasive ICP monitoring and its modalities will be set through a joint decision between neurosurgeons and intensive care physician, which will be led by clinical and instrumental data.

This study will be carried out in Intensive Care Unit and in Neurosurgery department.

Sample size assessment:

Sample size assessment has been performed by Monte Carlo simulation (B=500). Assuming a timing decrease (T2-T1) of 20 minutes in the procedure carried out by an intensivist compared to a neurosurgeon, with a mean time of 100 minutes, a standard deviation between center and intra-center of 10 minutes, 16 centers, each one with the same number of patients and a balance 1:1 between the two groups (intensivist:neurosurgeon), a total number of 64 patients (32 treated by intensivists and 32 by neurosurgeons), it allows us to evaluate the interest effect with a power of at least 95%, and a significance level of 5%.

This elevated power has been decided according to the simplicity of the assumed design (same number of entities and conditions for center) and not evaluable in his real configuration.

Statistical analysis plan:

Delta time in the placement of invasive ICP monitoring is assumed as T2-T1, declared in minutes.

Typology operator (neurosurgeon vs intensivist) impact on delta time will be evaluated through a multilevel model elaborated with a linear mixed model. The model will assume the center in which the maneuver is carried out as clustering factor. The place where the maneuver is carried out (intensive care unit vs operating room) and the confidence in performing the procedure (routine vs sporadic, defined as less than 5 times a year) will be assumed as covariates.

The incidence of complications, valued as a binary variable, will be evaluated through logistic model GLMM (generalized linear mixed model) with the organization exposed in the dedicated data element.

Timings are defined as:

* T0: suspect of pathology at risk for developing intracranial hypertension
* T1: neurointensive and neurosurgical indication to invasive ICP monitoring (it can be the time when brain CT is performed or, in the absence of a brain CT, the time at which indication to invasive ICP monitoring is stated)
* T2: skin incision at skull for BOLT/EVD placement

Place of positioning:

The place (intensive care unit or operating room) where the procedure is carried out must be declared.

ELIGIBILITY:
Inclusion Criteria:

* All patients with acute cerebral pathology with urgent indication to invasive intracranial pressure monitoring (intraparenchymal and intraventricular)
* Age greater than or equal to 18 years

Exclusion Criteria:

* Patients in whom indication to intraventricular catheter placement is stated for reasons other than the need of ICP monitoring (e.g. CSF drainage)
* Patients in whom indication to invasive intracranial pressure monitoring is not an urgent request
* Patients in whom a significative coagulation disorder is a contraindication for procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All acute brain Injured patients with urgent indication for invasive intracranial pressure monitoring
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-05-03 (Estimated); Study Completion 2022-05-03 (Estimated)

PRIMARY OUTCOMES:
To compare timing of invasive intracranial pressure monitoring performed by intensive care physicians and neurosurgeons | The time frame, will be from when the suspicion of a potential increase in ICP is given to when the actual skin incision for the insertion of the invasive catheter placement is performed. From indication up to 5 hours.
  The time frame, which also represents the main outcome of this study, is defined as the time-difference between the moment when indication of invasive ICP monitoring is given and the moment when the skin incision is performed for ICP monitoring placement.

SECONDARY OUTCOMES:
Comparative evaluation of post-procedural complications between intensivists and neurosurgeons | procedure to hospital discharge (in case of malfunction of the catheter, time is up to 12 hours after placement)
  Comparative evaluation of post-procedural complications (meningitis, catheter-placement related bleedings, wrong placement) between intensivists and neurosurgeons
Length of ICU stay | ICU admission to discharge, up to 30 days
  Length of ICU stay
length of hospital stay | hospital admission to discharge, up to 30 days
  length of hospital stay
duration of mechanical ventilation | from initiation of mechanical ventilation to weaning from the ventilator, up to 30 days.
  duration of mechanical ventilation
Glasgow Outcome Score at 3 months | 3 months after the acute event
  Glasgow Outcome Score

CONTACTS AND LOCATIONS:
Overall Officials: Frank Rasulo, Principal Investigator — Università degli Studi di Brescia
Locations (18):
- Italy (18):
  - Ospedale "M. Bufalini", Intensive Care Unit (U.O. Anestesia e Rianimazione), Neurosurgery Unit (U.O. Neurochirurgia), Cesena, Forlì-Cesena
  - Azienda Socio Sanitaria Territoriale Ovest Milanese (Neurosurgery Unit), Legnano, Milano
  - Ospedale Papa Giovanni XXIII, Intensive Care Unit (U.O. Anestesia e rianimazione 2), Neurosurgery Unit (U.O. Neurochirurgia), Bergamo
  - Spedali Civili di Brescia, Neurosurgery Unit (U.O. Neurochirugia), Brescia
  - Spedali Civili, Neuro Critical Care Unit (U.O. Anestesia e Rianimazione 2), Brescia
  - Azienda Ospedaliera Sant'Anna e San Sebastiano di Caserta (Neurosurgery Unit), Caserta
  - Ospedale Sant'Anna di Como, Intensive Care Unit (U.O. Anestesia e Rianimazione 2), Neurosurgery Unit (U.O. Neurochirurgia), Como
  - Ospedale Policlinico San Martino (Neurosurgery Unit), Genova
  - Ospedale Santa Maria Goretti (Neurosurgery Unit), Latina
  - Ospedale A. Manzoni (Intensive Care Unit and Neurosurgery Unit), Lecco
  - Ospedale Civile di Baggiovara (Neurosurgery Unit), Modena
  - Ospedale Santa Maria di Loreto Nuovo, Intensive Care Unit (U.O.C. di Terapia Intensiva e Rianimazione), Neurosurgery Unit (U.O.C. Neurochirurgia), Napoli
  - Azienda Ospedale Università Padova (Neurosurgery Unit), Padua
  - Policlinico San Matteo, Intensive Care Unit (U.O. Anestesia e rianimazione 2), Neurosurgery Unit (U.O. Neurochirurgia), Pavia
  - Policlinico Universitario Agostino Gemelli (Neurosurgery unit), Roma
  - Azienda Ospedaliera Città della Salute e della Scienza, Intensive Care Unit (U.O. Anestesia e Rianimazione), Neurosurgery Unit (U.O. Neurochirurgia), Torino
  - Presidio Ospedaliero Universitario Santa Maria della Misericordia, Intensive Care Unit (U.O. Anestesia e Rianimazione), Neurosurgery Unit, Udine
  - Azienda Ospedaliera Universitaria Integrata Verona (Neurosurgery Unit), Verona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Balestreri M, Czosnyka M, Hutchinson P, Steiner LA, Hiler M, Smielewski P, Pickard JD. Impact of intracranial pressure and cerebral perfusion pressure on severe disability and mortality after head injury. Neurocrit Care. 2006;4(1):8-13. doi: 10.1385/NCC:4:1:008. PMID 16498188
- [Background] Vik A, Nag T, Fredriksli OA, Skandsen T, Moen KG, Schirmer-Mikalsen K, Manley GT. Relationship of "dose" of intracranial hypertension to outcome in severe traumatic brain injury. J Neurosurg. 2008 Oct;109(4):678-84. doi: 10.3171/JNS/2008/109/10/0678. PMID 18826355
- [Background] Sheth KN, Stein DM, Aarabi B, Hu P, Kufera JA, Scalea TM, Hanley DF. Intracranial pressure dose and outcome in traumatic brain injury. Neurocrit Care. 2013 Feb;18(1):26-32. doi: 10.1007/s12028-012-9780-3. PMID 23055087
- [Background] Ko K, Conforti A. Training protocol for intracranial pressure monitor placement by nonneurosurgeons: 5-year experience. J Trauma. 2003 Sep;55(3):480-3; discussion 483-4. doi: 10.1097/01.TA.0000074111.04885.28. PMID 14501890
- [Background] Ehtisham A, Taylor S, Bayless L, Klein MW, Janzen JM. Placement of external ventricular drains and intracranial pressure monitors by neurointensivists. Neurocrit Care. 2009;10(2):241-7. doi: 10.1007/s12028-008-9097-4. PMID 18449808
- [Background] Barber MA, Helmer SD, Morgan JT, Haan JM. Placement of intracranial pressure monitors by non-neurosurgeons: excellent outcomes can be achieved. J Trauma Acute Care Surg. 2012 Sep;73(3):558-63; discussion 563-5. doi: 10.1097/TA.0b013e318265cb75. PMID 22929484
- [Background] Sadaka F, Kasal J, Lakshmanan R, Palagiri A. Placement of intracranial pressure monitors by neurointensivists: case series and a systematic review. Brain Inj. 2013;27(5):600-4. doi: 10.3109/02699052.2013.772238. Epub 2013 Mar 8. PMID 23473439

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT05045105/Prot_SAP_000.pdf